CLINICAL TRIAL: NCT05864456
Title: Evaluation of the Safety and Efficacy of the Prizvalve Pro™ Transcatheter Aortic Valve System in the Treatment of Patients With Severe Aortic Valve Stenosis Disease at High Surgical Risk
Brief Title: Prizvalve Pro™ Transcatheter Aortic Valve Replacement Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Collaborators: The General Hospital of Northern Theater Command (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prizvalve Pro-2023
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter aortic valve replacement (Experimental): Transcatheter aortic valve replacement with Prizvalve Pro™ transcatheter aortic valve system
  Interventions: Device: Prizvalve Pro™ transcatheter aortic valve system

INTERVENTIONS:
Device: Prizvalve Pro™ transcatheter aortic valve system — Transcatheter Aortic Valve Replacement

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of the Prizvalve Pro™ transcatheter aortic valve system in the treatment of patients with severe aortic stenosis who are at high risk of surgery or who are not suitable for surgery.

DETAILED DESCRIPTION:
This study is a multicenter, single-arm, prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years ;
2. Patients with symptomatic severe aortic valve stenosis (evaluated by echocardiography: transaortic valve pressure gradient ≥40mmHg (1mmHg=0.133kPa), or transaortic valve blood flow rate ≥4m/s, or aortic Valve area<1.0cm², or AVA <0.5cm² /m²);
3. Cardiac function NYHA ≥ II;
4. Life expectancy> 12 months;
5. Patients who are anatomically suitable for transcatheter aortic valve implantation;
6. Patients who have been evaluated by two or more cardiovascular surgeons as unsuitable for conventional surgery; or patients who have refused conventional surgery after adequate communication from the surgeon and who are at high risk for conventional surgery;
7. Patients who can understand the purpose of the trial and volunteer to participate in, sign the informed consent form and are willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Acute myocardial infarction occurred within 1 month before this treatment;
2. Congenital unicuspid aortic valve;
3. Any therapeutic cardiac operation that is performed within 30 days of the index procedure (Previous PCI or implantation of a permanent pacemaker are not considered exclusion criteria);
4. Patients with other prosthetic heart valves, prosthetic rings already implanted in the heart, or severe mitral valve closure insufficiency (>3+);
5. Patients with hematologic disorders or abnormalities that make surgical treatment inappropriate;
6. Untreated severe coronary artery stenosis that requires revascularization;
7. Patients with hemodynamic or respiratory instability, requiring continuous mechanical heart assistance or mechanical ventilation;
8. Patients who need emergency surgery for any reason;
9. Patients with hypertrophic cardiomyopathy with obstruction;
10. Severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) <20%;
11. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
12. Patients with left ventricular outflow tract obstruction;
13. A history of acute peptic ulcer or upper gastrointestinal bleeding within 3 months;
14. Patients who are allergy or resistance to cobalt-chromium alloy, contrast agents and related components;
15. Patients who are unable to receive anticoagulation or antiplatelet therapy;
16. Cerebrovascular accident occurred within 3 months, not including transient ischemic attack;
17. Severe aortic diseases, including abdominal aortic or thoracic aortic aneurysm, etc;
18. Active infective endocarditis or other active infections;
19. Patients who have participated in clinical trials of other drugs or medical devices before enrollment and have not yet reached the primary outcome of research;
20. The investigator judged that patient with poor compliance and could not complete the study as required.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint event rate at 30 days | 30 days after procedure
  Composite endpoint event includes all-cause death, stroke, myocardial infarction, permanent pacemaker implantation, serious vascular and access-related complications, surgical intervention for aortic valve reoperation, valve-in-valve surgery.

SECONDARY OUTCOMES:
Device success rate | Immediately after procedure
  Device success is defined as
  1. The device enters the vascular approach, be transported, released and implanted successfully, and the delivery system is removed from the body successfully;
  2. The implanted valve achieves the desired efficacy (mean transvalvular pressure difference <20 mmHg or peak flow velocity <3 m/s in the aortic valve, no severe prosthetic aortic regurgitation or perivalvular leak).
Procedural success rate | Immediately after procedure
  Procedure success is defined as
  1. Implantation of ≤2 valves, with the implanted valves placed in the appropriate anatomic position;
  2. No intraoperative or immediate postoperative mortality;
  3. The intended purpose of the procedure was achieved without serious intraoperative complications (coronary occlusion, septal perforation, mitral valve damage or incompetence, pericardial tamponade, surgical termination, and open-heart surgical treatment for cardiac surgery).
Delivery system and component performance evaluation | Immediately after procedure
  Delivery system performance evaluation includes delivery, transvalve, release positioning, balloon filling and retrieval, visibility, and retrieval performance.
  (For each assessment: 1-4 points；1=excellent, 2=good, 3=fair, 4=poor).
Valve function | Immediately after procedure, 1 day of discharge, 30 days, 1 year
  Valve function includes aortic orifice area, transvalvular pressure difference, valvular regurgitation, and perivalvular leakage.
Improvement in cardiac function | 1 day of discharge, 30 days, 1-5 year
  Cardiac function is based on the New York Heart Association (NYHA) classification scheme.
Improvement in quality of life | 30 days, 1 year
  The SF-12 rating scale is used to assess quality of life.
Incidence of all-cause mortality | Immediately after procedure, 1 day of discharge, 30 days, 1-5 year
  Rate of all-cause mortality during the trial. All-cause mortality includes cardiovascular morality and non-cardiovascular morality.
Incidence of myocardial infarction | Immediately after procedure, 1 day of discharge, 30 days, 1-5 year
  Rate of patients with myocardial infarction during the trial.
Incidence of disabling stroke | 1 day of discharge, 30 days, 1-5 year
  Rate of patients with disabling stroke during the trial.
Incidence of permanent pacemaker implantation | 1 day of discharge, 30 days, 1-5 year
  Rate of patients with permanent pacemaker implantation during the trial.
Incidence of serious vascular and access-related complications | Immediately after procedure, 1 day of discharge, 30 days, 1-5 year
  Rate of patients with serious vascular and access-related complications during the trial.
Incidence of serious bleeding | 1 day of discharge, 30 days, 1-5 year
  Rate of patients with serious bleeding during the trial.
Incidence of acute kidney injury | 1 day of discharge, 30 days, 1-5 year
  Rate of patients with acute kidney injury during the trial.
Incidence of major cardiovascular and cerebrovascular adverse events | 1 day of discharge, 30 days, 1-5 year
  Incidence of MACCE during the trial. MACCE is defined as death, stroke, myocardial infarction, arrhythmia, conduction block, and aortic valve reoperation (interventional or surgical).
Incidence of other TAVI-related complications | Immediately after procedure, 1 day of discharge, 30 days, 1-5 year
  Rate of patients with other TAVI-related complications during the trial. Other TAVI-related complications include conversion to surgery, valve-in-valve implantation, accidental cardiopulmonary mechanical assistance, coronary occlusion, ventricular septal perforation, mitral valve damage or loss of function, pericardial tamponade, endocarditis, valvular thrombosis, valvular ectopic (migration, embolization, erroneous release), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Professor, Study Chair — Principal coordinating investigator; Mao Chen, Professor, Principal Investigator — coordinating investigator; Kai Xu, Professor, Study Director — coordinating investigator
Locations (1):
- Shanghai NewMed Medical Co., Ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No